CLINICAL TRIAL: NCT02986490
Title: Influence of Magnesium Variations (Serum and Intra-erythrocyte) on Markers of Cardiometabolic Risk in Long-term Prescription of Antipsychotic Drugs: a Prospective Cohort Study
Brief Title: Magnesium Variations and Cardiometabolic Risk in Patients With Antipsychotic Drugs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UF 9362; 2014-A00381-46 (Other: FRANCE: Agence Nationale de Sécurité des Médicaments)
Record Dates: First submitted 2016-07-08; First posted 2016-12-08 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-07

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Bipolar Disorder
Keywords: Mental disorders; Antipsychotic agents; Magnesium; Cardiovascular risk factor; Metabolic syndrome
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Bipolar Disorder; Mental Disorders; Metabolic Syndrome | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- patient with antipsychotic/neuroleptic (Other): Blood sample performed on patients requiring the establishment of treatment with antipsychotic / neuroleptic
  Interventions: Biological: Blood sample

INTERVENTIONS:
Biological: Blood sample — Blood sample

SUMMARY:
Background: Antipsychotics can induce metabolic disorders such as obesity, hyperglycemia, dyslipidemia or metabolic syndrome. It has been observed that treatment with antipsychotic could be accompanied by a decrease in the concentration of serum magnesium. Low serum concentrations of magnesium are potentially a risk factor of cardiac sudden death (Peacock, 2010). Hypotheses linking magnesium and pathogenesis of cardiovacuscular diseases are multiple. Also, it seems to exist a close relationship between magnesium and carbohydrate metabolism. Most studies on the subject have generally studied plasmatic magnesium.

Objective : Describe the relationship between changes in serum and intra-erythrocyte magnesium and cardiometabolic risk in patients innitiating an antipsychotic treatment. A secondary objective is to specify the frequency, magnitude and time to onset of changes in plasma of magnesium levels under antipsychotic treatment.

Methods : This is a pilot single-center prospective cohort. After inclusion, patients status (including magnesium levels) will be evaluated (1 and 3 months of treatment) and that status will define the exposure criterion. Included patients will be followed for 1 year during which cardiometabolic markers will be measured.

Population : patients who are more than 18 years old with schizophrenia schizoaffective disorder or bipolar disorder, naive to antipsychotic treatment or off for more than 3 months and requiring the introduction of antipsychotic drug therapy. Patients will be recruited during consultations and stays in care units of Adult Psychiatry Unit of Montpellier University Hospital.

Factor studied: serum and intra-erythrocytic magnesium levels at beginning and during the antipsychotic treatment measured by a unique analyzer center. Changes in levels of hypomagnesemia expected during the treatment will determine exposure groups.

Outcome: cardiometabolic risk markers measured at the beginning and during the treatment will be fasting blood glucose, fasting plasma insulin, HOMA-IR [Ins (uU / mL) x Gly (mmol / L) / 22.5], lipid profile (total cholesterol, LDL, HDL), BMI, waist circumference and ECG (QTc).

Cofactors: age, sex, personal and family medical history, blood pressure, smoking, diet, physical activity, psychiatric disease, Global Impressions, anti-psychotic treatment and comedications.

Perspectives : to show that decreased in magnesium levels observed among patients starting antipsychotic treatment is associated with deterioration of cardiometabolic risk markers. The demonstration of this association could explain at least part the increased cardiovascular risk observed in this population. In the longer term, the results of this study would argue the implementation of an intervention research project studying magnesium supplementation to minimize the metabolic effects of antipsychotic medications.

DETAILED DESCRIPTION:
This is a pilot single-center prospective cohort. After inclusion, patients status (including magnesium levels) will be evaluated (1 and 3 months of treatment) and that status will define the exposure criterion. Included patients will be followed for 1 year during which cardiometabolic markers will be measured.

Patients will be recruited during consultations and stays in care units of Adult Psychiatry Unit of Montpellier University Hospital.

ELIGIBILITY:
Inclusion criteria:

* Patient with severe mental illness (schizophrenia and other disorders chronic psychotic, schizoaffective disorder and bipolar disorder.
* Patient naive to antipsychotic treatment or stopped for more than 3 months (more than 6 months for antipsychotic action extended) and requiring the introduction of antipsychotic therapy
* Patient informed and accepting the proposed follow-up (himself or his/her legal representative)
* Patient available for one year monitoring
* Patient affiliated or beneficiary of a social security insurance

Exclusion criteria:

* patient's opposition
* Pregnant or breastfeeding patient
* Patients on anti-psychotic or treatment stopped for less than 3 months (6 months for antipsychotic prolonged action)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-09; Primary Completion 2017-01 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with changes from baseline cardiometabolic risk | At 12 months
  Changes from baseline cardiometabolic risk is defined the following composite outcome : 15% increase in fasting plasma glucose and/or 15% increase in plasma fasting insulin and/or 15% increase in HOMA-IR [Ins (uU / mL) x Gly (mmol / L) / 22.5] and/or 15% increase in total cholesterol levels, or LDL-cholesterol and/or reduction of 15% of HDL-cholesterol and/or 2 points increased in BMI and/or increase of 5 cm in waist circumference and/or 10 msec increase in the QTc interval of the ECG.

SECONDARY OUTCOMES:
Proportion of patients with changes from baseline cardiometabolic risk | At 3 months
Proportion of patients with changes from baseline cardiometabolic risk | At 6 months
Proportion of patients with 15% increase in fasting plasma glucose | From baseline at 12 months
Proportion of patients with 15% increase in plasma fasting insulin | From baseline at 12 months
Proportion of patients with 15% increase in HOMA-IR [Ins (uU / mL) x Gly (mmol / L) / 22.5] | From baseline at 12 months
Proportion of patients with 15% increase in total cholesterol levels, or LDL-cholesterol and/or reduction of 15% of HDL-cholesterol | From baseline at 12 months
Proportion of patients with 2 points increased in BMI and/or increase of 5 cm in waist circumference | From baseline at 12 months
9. Proportion of patients with 10 msec increase in the QTc interval of the ECG | From baseline at 12 months
Change in zincemia | From baseline at 12 months
Change in zincemia | From baseline at 3 months
Change in zincemia | From baseline at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc FAILLIE, MD PhD, Principal Investigator — Montpellier University Hospital
Locations (1):
- Montpellier, France

IPD SHARING:
Plan to Share IPD: No